CLINICAL TRIAL: NCT07246122
Title: MRI-Guided Dynamic Support System for Scoliosis Correction (MRI-DSS)
Brief Title: MRI-Guided Dynamic Support System for Scoliosis Correction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20230614001
Record Dates: First submitted 2025-07-29; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: MRI; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AIS bracing group (Experimental): Moderate AIS patients wearing customized MRI compatible soft brace, supine position lie in the MRI device
  Interventions: Device: MRI-guided Dynamic Support System

INTERVENTIONS:
Device: MRI-guided Dynamic Support System — MRI-compatible pneumatic support system with customized padding inserted into the brace, used for image-guided adjustment of corrective pressure during MRI scanning

SUMMARY:
This prospective pilot study evaluates the feasibility and effectiveness of an MRI-guided dynamic support system (MRI-DSS) for rapid, quantitative correction of adolescent idiopathic scoliosis (AIS). The system uses MRI-compatible air padding supports and programmable pneumatic control to apply and adjust corrective forces in real time. AIS patients underwent MRI-guided bracing, with Cobb angles and biomechanical parameters measured at each pressure level.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10-16 years
* Diagnosis: Adolescent idiopathic scoliosis (Cobb angle 10-25°)
* No prior spinal surgery or other orthopedic conditions
* Able to provide informed consent
* Risser sign 0-5

Exclusion Criteria:

* Age <10 or >16 years
* Cobb angle <10° or >25°
* History of spinal surgery or other spine disorders
* Contraindications to MRI

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cobb angle | baseline
  degrees measured by MRI
Time to achieve target correction | immediately after the intervention
  measured in minutes

SECONDARY OUTCOMES:
Contact area and force distribution | immediately after the intervention
  measured by 3D MRI reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Chinese University of Hong Kong; Joanne Yip, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Tsim Sha Tsui, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No